CLINICAL TRIAL: NCT02436083
Title: The Value of Perioperative Antibiotics on the Success of Oral Free Flap Reconstructions
Brief Title: Antibiotics in Free Flaps Reconstructions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, thomas.muecke, responsible consultant, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MKG-2007
Record Dates: First submitted 2015-03-09; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Infection
MeSH Terms: interventions — Anti-Bacterial Agents; Cefuroxime

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): no antibiotics
- experimental group (Active Comparator): drug administration (antibiotic)
  Interventions: Drug: antibiotic (use of penicilline, unacid, cefuroxime)

INTERVENTIONS:
Drug: antibiotic (use of penicilline, unacid, cefuroxime) — prophylactic antibiotics
  Other Names: use of penicilline, unacid, cefuroxime
  Arms: experimental group

SUMMARY:
The purpose of this study is to monitor and compare peri-operative problems and outcomes of reconstructive surgery with microvascular free flaps in the head and neck region between groups of patients treated with perioperative antibiotics and a group of patients without antibiotics.

DETAILED DESCRIPTION:
Study Design and Patient Recruitment All clinical investigations have been conducted according to the principles expressed in the Declaration of Helsinki. Patient consent was written. Any patient who required reconstructive surgery for oncological reasons within the oral cavity with microvascular free flaps was eligible. Patients receiving preoperative neoadjuvant or previous adjuvant radiation therapy in their medical history were not included in this study as the protocols available are not comparable in doses and effect on the irradiated tissue.14 A prospective study was initiated from July of 2007 to June 2012. All patients were prospectively evaluated.

Postoperative Care The investigators standard regimen was to keep the patient sedated for one night on the intensive care unit and then transfer to the surgical ward. The specific intravenous antibiotic therapy was started 30 minutes before the operation and administered for 10 days.

Data Analysis Recorded parameters included: age, sex, preoperative medical history, American society of Anesthesiologists classification of preoperative status 15, diagnosis, stage of disease, defect localisation, type of microvascular free flap, choice of recipient vessels, flap success, rate and number of operative revisions, primary or secondary reconstruction, type of previous treatment (radiation or surgery), type of previous neck dissection (if any), microvascular complications, the total operative time, wound healing disturbances subdivided into dehiscence and infection at the neck, region of reconstruction, or donor site, and prophylactic antibiotic agent, if used. Infection was defined as a purulent discharge at the wounds.

Descriptive statistics for quantitative variables are given as the mean ± standard deviation. The data were analyzed with the "Statistical Package for the Social Sciences" software (IBM® SPSS® Statistics for Windows, Version 22.0; IBM Corp., Armonk, NY, USA). Figures are generated with SPSS and Microsoft® Office Excel (Microsoft Excel for Windows, release 11.0, 2003, Microsoft Corporation, Redmond, WA, USA). Multiple linear regression analyses were used to determine factors independently associated with the dependent variable wound infection or wound healing disturbances. 95% confidence intervals (95% CI) are also given. Differences were considered to be statistically significant for a two-sided p-value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who required reconstructive surgery for oncological reasons within the oral cavity with microvascular free flaps.

Exclusion Criteria:

* Healthy humans.
* Patients receiving preoperative neoadjuvant or previous adjuvant radiation therapy in their medical history.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Frequencies of wound infection detected by clinical examinations (daily for 2 weeks, 2 times per week afterwards) | participants will be followed for the duration of hospital stay (2 weeks) and a total of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denys J Loeffelbein, MD, DDS, PhD, Study Chair — Department of Oral and Maxillofacial Surgery

REFERENCES:
- [Derived] Mucke T, Rohleder NH, Rau A, Ritschl LM, Kesting M, Wolff KD, Mitchell DA, Loeffelbein DJ. The value of perioperative antibiotics on the success of oral free flap reconstructions. Microsurgery. 2015 Oct;35(7):507-11. doi: 10.1002/micr.22470. Epub 2015 Aug 7. PMID 26251066